CLINICAL TRIAL: NCT06732440
Title: Subthreshold Vestibular Stimulation as a Strategy for Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2004550; 4R00DC020759-02 (NIH)
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2024-12

CONDITIONS: Vestibular Hypofunction; Bilateral Vestibular Hypofunction; Presbyvestibulopathy; Healthy Controls
Keywords: Bilateral Vestibular Hypofunction; Vestibular Rehabilitation

STUDY DESIGN:
Intervention Model Description: Each participant will complete all four days of the study.
Masking Description: All participants will complete all elements of the study. However, they will be blinded to the nature of each day of the study (i.e., will be unaware of participation in a "sham" vs. "motion" stimulus).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balance training performed with and without added subthreshold conditioning. (Experimental): Each participant in this single group design will complete the same three conditions of the experiment in a randomized order.
  Interventions: Behavioral: Subthreshold Vestibular Conditioning; Behavioral: Balance Training; Other: Balance Training Plus Subthreshold Conditioning

INTERVENTIONS:
Behavioral: Subthreshold Vestibular Conditioning — Subthreshold vestibular conditioning will be performed while seated on a motion platform and blindfolded. The stimulus will consist of a pseudorandom sum-of-sinusoids roll tilt motion (~0.08 to 1 Hz) delivered at a peak velocity equal to 57.4% of the measured baseline roll tilt perceptual threshold (e.g., 0.574°/s for a 1 °/s threshold). The participant will be informed that while the chair may vibrate or move slightly, the motion will not occur in any particular direction.
Behavioral: Balance Training — Balance training will consist of progressive exposure to continuous one-dimensional roll pseudorandom platform perturbations delivered using a 6DoF motion platform. Participants will stand on a MOOG hexapod motion platform and will be secured using a safety harness tethered to the ceiling and a full enclosure of safety rails. Roll tilt perturbations will be progressed by gradually increasing the displacement/velocity/acceleration of the platform motion.
Other: Balance Training Plus Subthreshold Conditioning — Subthreshold vestibular conditioning will be performed while seated on a motion platform and blindfolded prior to each bout of balance training. Subthreshold conditioning will consist of a pseudorandom sum-of-sinusoids roll tilt motion (~0.08 to 1 Hz) delivered at a peak velocity equal to 57.4% of the measured baseline roll tilt perceptual threshold (e.g., 0.574°/s for a 1 °/s threshold). The participant will be informed that while the chair may vibrate or move slightly, the motion will not occur in any particular direction. Balance training will consist of progressive exposure to continuous two-dimensional (2D) pseudorandom platform perturbations delivered using a 6DoF motion platform. 2D perturbations (roll and pitch tilt) will be progressed by gradually increasing the displacement/velocity/acceleration of the motion stimulus.

SUMMARY:
The nervous system responds to changes in external or internal conditions by altering the behavior of neurons through multiple forms of neural plasticity. A specific form of plasticity, "homeostatic plasticity", stabilizes neural activity by driving the excitability of neurons toward a "set-point" level of activity. Over the last six years, new data have come to light showing that the vestibular system also possess a robust capacity to modulate sensitivity to self-motion cues in response to prolonged periods of motion. Collectively, these studies have demonstrated a capacity to use motion perturbations (i.e., low, or high levels of vestibular stimulation) to dynamically adjust the sensitivity of the vestibular system on both the single neuron and behavioral levels. The ability to use subthreshold motion stimuli to drive plasticity in the vestibular system motivates this study. The investigators aim to determine the impact of subthreshold motion on (a) balance performance and (b) balance training in individuals with peripheral vestibular hypofunction.

DETAILED DESCRIPTION:
The investigators aim to test (1) if sub threshold motion improves motion perception, (2) if sub threshold motion improves balance performance, and (3) if sub threshold motion prior to balance training leads to improved balance performance. Twenty-four subjects with peripheral vestibular hypofunction (12 with bilateral and 12 with unilateral hypofunction) and twenty-four healthy control participants will complete the study. Each participant will complete four visits to the laboratory. Day 1 will measure the capacity to modify balance and self-motion perception after a single block of subthreshold motion, including any retention effects after a washout period. Days 2-4 will be performed in random order and will test changes in balance and self-motion perception after (a) repeated balance training, (b) repeated subthreshold motion, and (c) balance training combined with sub threshold motion.

ELIGIBILITY:
Inclusion Criteria for Bilateral Vestibular Hypofunction:

1. Bilateral lateral canal VOR gain of < 0.8 on video head impulse testing OR bilateral positive bedside head impulse test

Inclusion Criteria for Unilateral Vestibular Hypofunction:

1. Unilateral yaw aVOR gain of < 0.8 on video head impulse testing OR unilateral positive bedside head impulse test

Inclusion Criteria for all Participants:

1. Must be able to stand for 5 minutes unassisted
2. No leg or foot amputations
3. No lower limb braces
4. Not currently pregnant by self-report
5. Weight <= 300 pounds (due to limitations of testing equipment)

Exclusion Criteria for all participants:

1. Severe head trauma or traumatic brain injury
2. History of seizures
3. Alternative neurologic illness or condition known to impact vestibular or balance function (e.g., stroke, neurodegenerative disorders, demyelinating illness)
4. Major psychiatric (e.g., panic disorder, psychosis, etc.) disorder
5. Any of the following eye diseases or conditions: amblyopia (or "lazy eye") or history of amblyopia, diagnosis of age- related macular degeneration, retina dystrophy, glaucoma, cataracts,
6. Recent (<6 months) orthopedic injury that may affect test performance
7. Recent surgery (< 6 months) that may impact test performance.
8. Other severe health problems (heart disease, pulmonary disease, cancer, etc.) that may affect test performance
9. Due to potentially nauseogenic nature of some motions and to protect fetus and mother, pregnant women will also be excluded from this study

   * Since the investigators cannot address every possible potential individual recruit in advance, additional exclusion criteria may be required.

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Perturbed Stance Postural Control | At each of the 4 visits, outcome measures will be captured at (1) beginning of the visit (i.e., baseline), (2) post-intervention (20 minutes after baseline), and (3) post-washout (20 minutes after the post-intervention assessment).
  The RMSD of mediolateral (ML) and anteroposterior (AP) postural sway will be measured in response to pseudorandom two-dimensional mediolateral and anteroposterior tilts of the support surface delivered using a 6DoF motion platform. Participants will stand with eyes closed and feet at a standardized distance on top of the motion platform. The platform will tilt simultaneously in both the roll and pitch planes, with each plane of tilt having independent frequency spectra (~0.08 to 1 Hz). The perturbation test will last approximately 2 minutes.
Vestibular Perceptual Thresholds - 0.5Hz Roll Tilt | At each of the 4 visits, outcome measures will be captured at (1) beginning of the visit (i.e., baseline), (2) post-intervention (20 minutes after baseline), and (3) post-washout (20 minutes after the post-intervention assessment).
  Vestibular perceptual thresholds will be measured using a forced-choice direction recognition task using methods that the investigators have used extensively. Subjects will be tilted in the coronal plane (i.e., roll tilt) in one of two directions (e.g., towards the left or right) in complete darkness while seated on a 6DoF platform. To mask potential auditory directionality cues, auditory "noise" - uncorrelated with motion (amplitude, direction, or type) - will be applied at approximately 60 dB SPL. Motion stimuli will consist of single cycles of sinusoidal acceleration. After each motion, the participant will be asked to judge the direction of the tilt stimulus, with the threshold being defined as the smallest velocity of tilt that can be accurately perceived.

OTHER OUTCOMES:
Symptom Severity | Subjective outcome measures will be captured only on the first visit, prior to completing any intervention conditions.
  Each participant will complete standardized questionnaires to assess symptom severity including: (a) dizziness (Dizziness Handicap Inventory), a measure of perceived handicap due to dizziness, with higher scores indicating more severe disability related handicap; (b) balance confidence (Activities Balance Confidence Scale), a measure of balance confidence, with higher scores indicating a higher degree of confidence in balance; and (c) impact of vestibular symptoms on daily life (Vestibular Activities of Daily Living Scale), a measure describing the impact of vestibular symptoms on activities of daily living, with higher scores indicating a greater impact of vestibular symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton University, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wagner AR, Kobel MJ, Tajino J, Merfeld DM. Improving self-motion perception and balance through roll tilt perceptual training. J Neurophysiol. 2022 Sep 1;128(3):619-633. doi: 10.1152/jn.00092.2022. Epub 2022 Jul 27. PMID 35894439
- [Background] Dietrich H, Straka H. Prolonged vestibular stimulation induces homeostatic plasticity of the vestibulo-ocular reflex in larval Xenopus laevis. Eur J Neurosci. 2016 Jul;44(1):1787-96. doi: 10.1111/ejn.13269. Epub 2016 Jun 1. PMID 27152983
- [Background] Kobel MJ, Wagner AR, Merfeld DM, Mattingly JK. Vestibular Thresholds: A Review of Advances and Challenges in Clinical Applications. Front Neurol. 2021 Feb 19;12:643634. doi: 10.3389/fneur.2021.643634. eCollection 2021. PMID 33679594